CLINICAL TRIAL: NCT01470664
Title: A Proof-of-Concept, Multi-center, Randomized, Double-Masked Study to Evaluate the Clinical Efficacy and Safety of FST-100 Ophthalmic Suspension in the Treatment of Acute Adenoviral Conjunctivitis
Brief Title: FST-100 in the Treatment of Acute Adenoviral Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FST100-AVC-004
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Acute Adenoviral Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- FST-100 (Experimental)
  Interventions: Drug: FST-100
- FST-100 (Component #1) (Experimental)
  Interventions: Drug: FST-100 (Component #1)
- FST-100 Vehicle (Placebo Comparator)
  Interventions: Drug: FST-100 Vehicle

INTERVENTIONS:
Drug: FST-100 — 0.1% dexamethasone and 0.6% polyvinylpyrrolidone iodine (PVP-Iodine)
  Arms: FST-100
Drug: FST-100 (Component #1) — 0.6% PVP-Iodine ophthalmic solution alone
  Arms: FST-100 (Component #1)
Drug: FST-100 Vehicle — FST-100 Vehicle
  Arms: FST-100 Vehicle

SUMMARY:
This randomized, double masked, multi-center study is being conducted to support the safety and efficacy of FST-100 for the treatment of acute adenoviral conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of suspected acute adenoviral conjunctivitis in at least one eye.

Exclusion Criteria:

* Have a known sensitivity to any of the components of FST-100 or FST-100 vehicle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2012-12-17 (Actual); Primary Completion 2014-05-23 (Actual); Study Completion 2014-05-23 (Actual)

PRIMARY OUTCOMES:
Adenoviral eradication and clinical resolution of the infection | 6-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Ora, Inc., Andover, Massachusetts, United States
- Ora, Inc., Noida, India